CLINICAL TRIAL: NCT02932085
Title: Pilot Study for the Effects of Transcranial Magnetic Stimulation on the Brain Using an Electronic Medical Device: A Single Institution, Randomized, Double-blind, Sham-controlled Study Using Multimodal Neuroimaging in Healthy Young Adults
Brief Title: Pilot Study for the Effects of Transcranial Magnetic Stimulation on the Brain Using an Electronic Medical Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Sujung Yoon, Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NRF_rTMS
Record Dates: First submitted 2016-09-26; First posted 2016-10-13 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Transcranial magnetic stimulation; Magnetic resonance imaging; Magnetic resonance spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS + Wash-out period + Sham (Active Comparator): * Five consecutive daily repetitive transcranial magnetic stimulation sessions (Neurostar TMS Therapy System, NeuroStar XPLOR System)
  * Two weeks wash-out period
  * Five consecutive daily sham stimulation sessions
  Interventions: Device: Neurostar TMS Therapy System, NeuroStar XPLOR System
- Sham + Wash-out period + rTMS (Sham Comparator): * Five consecutive daily sham stimulation sessions (Neurostar TMS Therapy System, NeuroStar XPLOR System)
  * Two weeks wash-out period
  * Five consecutive daily repetitive transcranial magnetic stimulation sessions
  Interventions: Device: Neurostar TMS Therapy System, NeuroStar XPLOR System

INTERVENTIONS:
Device: Neurostar TMS Therapy System, NeuroStar XPLOR System — Repetitive transcranial magnetic stimulation

SUMMARY:
This study is a randomized, double-blind, and sham-controlled trial to examine the effects of transcranial magnetic stimulation on the brain of health individuals.

DETAILED DESCRIPTION:
The efficacy of repetitive transcranial magnetic stimulation on the brain will be assessed by multimodal neuroimaging in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19-39 years
* Informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* High fever patient
* Current and past history of seizure or epilepsy
* Evidence of epilepsy on EEG
* Pregnancy or possibility of pregnancy during period
* Major medical or neurological illnesses
* Evidence of alcohol intake on alcohol breath test
* Contraindications to MRI scans and transcranial magnetic stimulation
* Risk of skin burns
* Use of medications that could have influenced on the study

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Metabolic brain changes in magnetic resonance imaging by computational approaches | after 5 sessions (1 session/day) equals 5 days

SECONDARY OUTCOMES:
Functional brain changes in magnetic resonance imaging by computational approaches | after 5 sessions (1 session/day) equals 5 days
Standardized scores on a neuropsychological test battery | after 5 sessions (1 session/day) equals 5 days
Analysis of EEG activity | after 5 sessions (1 session/day) equals 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong H, Kim RY, Song Y, Suh C, Lee H, Lyoo IK, Yoon S, Lim SM, Lee S. Genetic profile for dopamine signaling predicts brain functional reactivity to repetitive transcranial magnetic stimulation. Eur Arch Psychiatry Clin Neurosci. 2023 Feb;273(1):99-111. doi: 10.1007/s00406-022-01436-2. Epub 2022 Aug 11. PMID 35951113